CLINICAL TRIAL: NCT04263207
Title: Observational Study for the Evaluation of the Role of HIV-1 Tat Protein and Anti-Tat Immune Response in Peripheral Blood HIV Reservoir Dynamics
Brief Title: Observational Study for the Evaluation of the Role of HIV-1 Tat Protein and Anti-Tat Immune Response In HIV Reservoir
Acronym: ISS OBS T-005
Status: Suspended | Type: Observational
Why Stopped: Study halted prematurely due to the difficulties in dedicating the human resources necessary to conduct the study deriving from the COVID-19 pandemic, but potentially will resume
Sponsor: Barbara Ensoli, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, Director, National HIV/AIDS Research Center (CNAIDS), Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: ISS OBS T-005
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Immune responses; Tat; HIV reservoire; Biomarkers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Periferal blood mononuclear cells and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anti-Tat Ab positive subjects
  Interventions: Other: No intervention
- anti-Tat Ab negative subjects
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A longitudinal observational study in HIV-infected subjects receiving cART addressed to explore the effect of the Tat protein and anti-Tat immunity on the formation and maintenance of HIV-1 virus reservoir.

DETAILED DESCRIPTION:
The study is designed as a longitudinal observational study addressed to identify the effects of Tat protein and humoral/cellular anti-Tat immune responses (induced in the natural infection or by Tat vaccination) in HIV-1 reservoir dynamics in blood of HIV infected patients receiving cART. HIV DNA data will be used for analyzing the decay dynamics.

The primary objective of the study is to determine the rate of decay of total HIV DNA in blood of anti-Tat antibody (Ab) positive versus anti-Tat Ab negative HIV patients receiving cART.

The secondary objectives of the study are to relate the HIV DNA decay data to:

1. the persistence of anti-Tat humoral responses;
2. biomarkers of HIV reservoir stability potentially affected by the Tat protein or anti-Tat immune responses, including: i) apoptotic/survival index of CD4+ T cells; ii) reactivation dynamics of latent HIV in resting CD4+ T cells upon exposure to Tat protein and/or activation stimuli; iii) cellular and humoral biomarkers relevant to inflammation and immune dysregulation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosis of HIV-1 infection
3. To be under cART treatment
4. CD4+ T-cell count ≥250 cells/microliters
5. Testing for anti-Tat Ab performed during pre-screening
6. Signed informed consent

Exclusion Criteria:

1. Current therapy with immunomodulators or immunosuppressive drugs or chemotherapy for neoplastic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected adult subjects of either gender, ≥18 years old, under cART, with CD4+ T-cell count ≥250 cells/µL.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
HIV proviral DNA levels | Baseline and through study completion, an average of 3 years
  Changes of total HIV-1 proviral DNA copies/1.000.000 CD4+ T-cells
HIV plasma viremia | Baseline and through study completion, an average of 3 years
  Changes of HIV plasma viral load (copies/mL)
CD4+ and CD8+ T-cell levels | Baseline and through study completion, an average of 3 years
  Changes of CD4+ and CD8+ T-cell counts (cells/microL)

SECONDARY OUTCOMES:
lymphocytes subset apoptosis | Baseline and through study completion, an average of 3 years
  Apoptotic index of isolated lymphocytes subsets
Induction of replication of competent latent HIV-1 from resting CD4+ T-cell | Baseline and through study completion, an average of 3 years
  Quantification of replication competent latent HIV-1 from isolated resting CD4+ T cells [TZM-bl cell based assay (TZA)]
Inflammation/immune activation biomarkers | Baseline and through study completion, an average of 3 years
  Plasma levels of inflammation and immune activation biomarkers
Anti-Tat Ab isotypes | Baseline and through study completion, an average of 3 years
  Anti-Tat humoral response in terms of anti-Tat IgM, IgG and IgA Ab

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Dermatology STI Unit San Gallicano Dermatologic Institute , IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murray AJ, Kwon KJ, Farber DL, Siliciano RF. The Latent Reservoir for HIV-1: How Immunologic Memory and Clonal Expansion Contribute to HIV-1 Persistence. J Immunol. 2016 Jul 15;197(2):407-17. doi: 10.4049/jimmunol.1600343. PMID 27382129
- [Background] Avettand-Fenoel V, Hocqueloux L, Ghosn J, Cheret A, Frange P, Melard A, Viard JP, Rouzioux C. Total HIV-1 DNA, a Marker of Viral Reservoir Dynamics with Clinical Implications. Clin Microbiol Rev. 2016 Oct;29(4):859-80. doi: 10.1128/CMR.00015-16. PMID 27559075
- [Background] Blankson JN, Finzi D, Pierson TC, Sabundayo BP, Chadwick K, Margolick JB, Quinn TC, Siliciano RF. Biphasic decay of latently infected CD4+ T cells in acute human immunodeficiency virus type 1 infection. J Infect Dis. 2000 Dec;182(6):1636-42. doi: 10.1086/317615. Epub 2000 Nov 8. PMID 11069234
- [Background] Siliciano JM, Siliciano RF. The Remarkable Stability of the Latent Reservoir for HIV-1 in Resting Memory CD4+ T Cells. J Infect Dis. 2015 Nov 1;212(9):1345-7. doi: 10.1093/infdis/jiv219. Epub 2015 Apr 15. No abstract available. PMID 25877551
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Sigal A, Kim JT, Balazs AB, Dekel E, Mayo A, Milo R, Baltimore D. Cell-to-cell spread of HIV permits ongoing replication despite antiretroviral therapy. Nature. 2011 Aug 17;477(7362):95-8. doi: 10.1038/nature10347. PMID 21849975
- [Background] Lorenzo-Redondo R, Fryer HR, Bedford T, Kim EY, Archer J, Pond SLK, Chung YS, Penugonda S, Chipman J, Fletcher CV, Schacker TW, Malim MH, Rambaut A, Haase AT, McLean AR, Wolinsky SM. Persistent HIV-1 replication maintains the tissue reservoir during therapy. Nature. 2016 Feb 4;530(7588):51-56. doi: 10.1038/nature16933. Epub 2016 Jan 27. PMID 26814962
- [Background] Deng K, Pertea M, Rongvaux A, Wang L, Durand CM, Ghiaur G, Lai J, McHugh HL, Hao H, Zhang H, Margolick JB, Gurer C, Murphy AJ, Valenzuela DM, Yancopoulos GD, Deeks SG, Strowig T, Kumar P, Siliciano JD, Salzberg SL, Flavell RA, Shan L, Siliciano RF. Broad CTL response is required to clear latent HIV-1 due to dominance of escape mutations. Nature. 2015 Jan 15;517(7534):381-5. doi: 10.1038/nature14053. Epub 2015 Jan 7. PMID 25561180
- [Background] Hosmane NN, Kwon KJ, Bruner KM, Capoferri AA, Beg S, Rosenbloom DI, Keele BF, Ho YC, Siliciano JD, Siliciano RF. Proliferation of latently infected CD4+ T cells carrying replication-competent HIV-1: Potential role in latent reservoir dynamics. J Exp Med. 2017 Apr 3;214(4):959-972. doi: 10.1084/jem.20170193. Epub 2017 Mar 24. PMID 28341641
- [Background] Jordan A, Defechereux P, Verdin E. The site of HIV-1 integration in the human genome determines basal transcriptional activity and response to Tat transactivation. EMBO J. 2001 Apr 2;20(7):1726-38. doi: 10.1093/emboj/20.7.1726. PMID 11285236
- [Background] C Quaresma AJ, Bugai A, Barboric M. Cracking the control of RNA polymerase II elongation by 7SK snRNP and P-TEFb. Nucleic Acids Res. 2016 Sep 19;44(16):7527-39. doi: 10.1093/nar/gkw585. Epub 2016 Jul 1. PMID 27369380
- [Background] Weinberger LS, Burnett JC, Toettcher JE, Arkin AP, Schaffer DV. Stochastic gene expression in a lentiviral positive-feedback loop: HIV-1 Tat fluctuations drive phenotypic diversity. Cell. 2005 Jul 29;122(2):169-82. doi: 10.1016/j.cell.2005.06.006. PMID 16051143
- [Background] Razooky BS, Pai A, Aull K, Rouzine IM, Weinberger LS. A hardwired HIV latency program. Cell. 2015 Feb 26;160(5):990-1001. doi: 10.1016/j.cell.2015.02.009. PMID 25723172
- [Background] Cafaro A, Sgadari C, Picconi O, Tripiciano A, Moretti S, Francavilla V, Pavone Cossut MR, Butto S, Cozzone G, Ensoli F, Monini P, Ensoli B. "cART intensification by the HIV-1 Tat B clade vaccine: progress to phase III efficacy studies". Expert Rev Vaccines. 2018 Feb;17(2):115-126. doi: 10.1080/14760584.2018.1418666. Epub 2017 Dec 22. PMID 29243498
- [Background] Frankel AD, Pabo CO. Cellular uptake of the tat protein from human immunodeficiency virus. Cell. 1988 Dec 23;55(6):1189-93. doi: 10.1016/0092-8674(88)90263-2. PMID 2849510
- [Background] Ensoli B, Buonaguro L, Barillari G, Fiorelli V, Gendelman R, Morgan RA, Wingfield P, Gallo RC. Release, uptake, and effects of extracellular human immunodeficiency virus type 1 Tat protein on cell growth and viral transactivation. J Virol. 1993 Jan;67(1):277-87. doi: 10.1128/JVI.67.1.277-287.1993. PMID 8416373
- [Background] Mousseau G, Kessing CF, Fromentin R, Trautmann L, Chomont N, Valente ST. The Tat Inhibitor Didehydro-Cortistatin A Prevents HIV-1 Reactivation from Latency. mBio. 2015 Jul 7;6(4):e00465. doi: 10.1128/mBio.00465-15. PMID 26152583
- [Background] Kessing CF, Nixon CC, Li C, Tsai P, Takata H, Mousseau G, Ho PT, Honeycutt JB, Fallahi M, Trautmann L, Garcia JV, Valente ST. In Vivo Suppression of HIV Rebound by Didehydro-Cortistatin A, a "Block-and-Lock" Strategy for HIV-1 Treatment. Cell Rep. 2017 Oct 17;21(3):600-611. doi: 10.1016/j.celrep.2017.09.080. PMID 29045830
- [Background] Johnson TP, Patel K, Johnson KR, Maric D, Calabresi PA, Hasbun R, Nath A. Induction of IL-17 and nonclassical T-cell activation by HIV-Tat protein. Proc Natl Acad Sci U S A. 2013 Aug 13;110(33):13588-93. doi: 10.1073/pnas.1308673110. Epub 2013 Jul 29. PMID 23898208
- [Background] Lopez-Huertas MR, Mateos E, Sanchez Del Cojo M, Gomez-Esquer F, Diaz-Gil G, Rodriguez-Mora S, Lopez JA, Calvo E, Lopez-Campos G, Alcami J, Coiras M. The presence of HIV-1 Tat protein second exon delays fas protein-mediated apoptosis in CD4+ T lymphocytes: a potential mechanism for persistent viral production. J Biol Chem. 2013 Mar 15;288(11):7626-7644. doi: 10.1074/jbc.M112.408294. Epub 2013 Jan 30. PMID 23364796
- [Background] Zauli G, Gibellini D, Caputo A, Bassini A, Negrini M, Monne M, Mazzoni M, Capitani S. The human immunodeficiency virus type-1 Tat protein upregulates Bcl-2 gene expression in Jurkat T-cell lines and primary peripheral blood mononuclear cells. Blood. 1995 Nov 15;86(10):3823-34. PMID 7579350
- [Background] Chiozzini C, Collacchi B, Nappi F, Bauer T, Arenaccio C, Tripiciano A, Longo O, Ensoli F, Cafaro A, Ensoli B, Federico M. Surface-bound Tat inhibits antigen-specific CD8+ T-cell activation in an integrin-dependent manner. AIDS. 2014 Sep 24;28(15):2189-200. doi: 10.1097/QAD.0000000000000389. PMID 25313583
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Ensoli B, Nchabeleng M, Ensoli F, Tripiciano A, Bellino S, Picconi O, Sgadari C, Longo O, Tavoschi L, Joffe D, Cafaro A, Francavilla V, Moretti S, Pavone Cossut MR, Collacchi B, Arancio A, Paniccia G, Casabianca A, Magnani M, Butto S, Levendal E, Ndimande JV, Asia B, Pillay Y, Garaci E, Monini P; SMU-MeCRU study group. HIV-Tat immunization induces cross-clade neutralizing antibodies and CD4(+) T cell increases in antiretroviral-treated South African volunteers: a randomized phase II clinical trial. Retrovirology. 2016 Jun 9;13(1):34. doi: 10.1186/s12977-016-0261-1. PMID 27277839
- [Background] Finzi D, Blankson J, Siliciano JD, Margolick JB, Chadwick K, Pierson T, Smith K, Lisziewicz J, Lori F, Flexner C, Quinn TC, Chaisson RE, Rosenberg E, Walker B, Gange S, Gallant J, Siliciano RF. Latent infection of CD4+ T cells provides a mechanism for lifelong persistence of HIV-1, even in patients on effective combination therapy. Nat Med. 1999 May;5(5):512-7. doi: 10.1038/8394. PMID 10229227
- [Background] Sanyal A, Mailliard RB, Rinaldo CR, Ratner D, Ding M, Chen Y, Zerbato JM, Giacobbi NS, Venkatachari NJ, Patterson BK, Chargin A, Sluis-Cremer N, Gupta P. Novel assay reveals a large, inducible, replication-competent HIV-1 reservoir in resting CD4+ T cells. Nat Med. 2017 Jul;23(7):885-889. doi: 10.1038/nm.4347. Epub 2017 May 29. PMID 28553933
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Background] Sgadari C, Barillari G, Palladino C, Bellino S, Taddeo B, Toschi E, Ensoli B. Fibroblast Growth Factor-2 and the HIV-1 Tat Protein Synergize in Promoting Bcl-2 Expression and Preventing Endothelial Cell Apoptosis: Implications for the Pathogenesis of AIDS-Associated Kaposi's Sarcoma. Int J Vasc Med. 2011;2011:452729. doi: 10.1155/2011/452729. Epub 2011 Oct 9. PMID 22007303
- [Background] Sgadari C, Monini P, Tripiciano A, Picconi O, Casabianca A, Orlandi C, Moretti S, Francavilla V, Arancio A, Paniccia G, Campagna M, Bellino S, Meschiari M, Nozza S, Sighinolfi L, Latini A, Muscatello A, Saracino A, Di Pietro M, Galli M, Cafaro A, Magnani M, Ensoli F, Ensoli B. Continued Decay of HIV Proviral DNA Upon Vaccination With HIV-1 Tat of Subjects on Long-Term ART: An 8-Year Follow-Up Study. Front Immunol. 2019 Feb 13;10:233. doi: 10.3389/fimmu.2019.00233. eCollection 2019. PMID 30815001
- [Background] Cafaro A, Tripiciano A, Picconi O, Sgadari C, Moretti S, Butto S, Monini P, Ensoli B. Anti-Tat Immunity in HIV-1 Infection: Effects of Naturally Occurring and Vaccine-Induced Antibodies Against Tat on the Course of the Disease. Vaccines (Basel). 2019 Aug 26;7(3):99. doi: 10.3390/vaccines7030099. PMID 31454973
- [Background] Moretti S, Cafaro A, Tripiciano A, Picconi O, Butto S, Ensoli F, Sgadari C, Monini P, Ensoli B. HIV therapeutic vaccines aimed at intensifying combination antiretroviral therapy. Expert Rev Vaccines. 2020 Jan;19(1):71-84. doi: 10.1080/14760584.2020.1712199. Epub 2020 Jan 19. PMID 31957513